CLINICAL TRIAL: NCT03173924
Title: Evaluation of 18F-DCFPyL PSMA- Versus 18F-NaF-PET Imaging for Detection of Metastatic Prostate Cancer
Brief Title: 18F-DCFPyL PSMA- Versus 18F-NaF-PET Imaging for Detection of Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 170089; 17-C-0089
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Metastatic Prostate Cancer; Prostatic Neoplasms; Prostate Cancer; Prostatic Cancer; Prostate Neoplasms
Keywords: Small Molecule; Radiolabeled; PSA; Diagnostic; PMSA
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Experimental intervention (Experimental): 18F-DCFPyL is administered to cohorts
  Interventions: Drug: 18F-NaF; Drug: 18F-DCFPyL; Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-NaF — Baseline IV followed by PET/CT IMAGING
Drug: 18F-DCFPyL — Baseline IV followed by PET/CT IMAGING. Additional 18F-DCFPyL PET/CTs might be performed during the subject s follow up period if, in the opinion of the referring clinician, there has been a considerable change in patient status (progression or response) based on clinical grounds/PSA value or to help assess changes of standard of care therapy.
Drug: 18F-FDG — Baseline IV followed by PET/CT IMAGING. Additional 18F-FDG PET/CTs may be obtained per PI discretion within a 21-day window relative to each 18F-DCFPyL PET/CTs.

SUMMARY:
Background:

Prostate cancer is the second leading cause of cancer deaths in American men. Few options exist to create images of this type of cancer. Researchers think an experimental radiotracer called 18F-DCFPyL could find sites of cancer in the body.

Objective:

To see if 18F-DCFPyL can identify sites of prostate cancer in people with the disease.

Eligibility:

People ages 18 and older who have metastatic prostate cancer

Design:

Participants will be screened with:

* Blood tests
* Physical exam
* Medical history

Participants will be assigned to 1 of 2 groups based on their PSA.

Participants will have 18F-DCFPyL injected into a vein. About 2 hours later they will have a whole-body Positron Emission

Tomography/Computed Tomography (PET/CT). For the scan, they will lie on their back on the scanner table while it takes pictures of the body. This lasts about 50 minutes.

On another day, participants will have 18F -NaF injected into a vein. About 1 hour later, they will have a whole-body PET/CT.

Participants will be contacted 1 3 days later for follow-up. They may undergo PET/Magnetic Resonance Imaging (MRI) either after having a 18F-DCFPyL PET/CT, or in place of PET/CT imaging. A tube may be placed in the rectum. More coils may be wrapped around the outside of the pelvis.

If the 18F-DCFPyL PET/CT is positive participants will be encouraged to undergo a biopsy of one of the tumors. The biopsy will be taken through a needle put through the skin into the tumor.

Participants will be followed for 1 year. During this time researchers will collect information about their prostate cancer, such as PSA levels and biopsy results.

About 4-6 months after scanning is completed, participants may have a tumor biopsy. The biopsy will be taken through a needle put through the skin into the tumor.

...

DETAILED DESCRIPTION:
Background:

The objective of this study is to evaluate a radiolabeled urea-based small molecule inhibitor of prostate-specific membrane antigen (PSMA), [18F] DCFPyL (DCFPyL) PET/CT (or PET/MRI imaging if available) for detection of metastatic prostate cancer

PSMA is a well characterized histological marker of prostate cancer tumor aggressiveness and metastatic potential

Our preliminary first-in-human studies demonstrate high specific uptake of a first generation less avid compound, DCFBC, in metastatic prostate cancer and demonstrated feasibility for prostate cancer metastatic detection.

We propose to assess the ability of DCFPyL PET to detect metastatic prostate cancer by visual qualitative and quantitative SUV analysis. Correlation will be made to sites of suspected bony metastatic disease detected by ultra-sensitive but less specific [18F] Sodium Fluoride (NaF)-PET/CT imaging and all sites of suspected disease detected by [18F] Fluorodeoxyglucose (FDG) for prostate cancer.

Objective:

To compare the diagnostic sensitivity of DCFPyL-PET/CT (or PET/MRI imaging if available) to NaF-PET/CT for detection of prostate cancer bone metastasis based on comparison to reference standard of care conventional imaging modalities (CIM); such as CT and whole body bone scintigraphy incorporating prior and follow-up scans and histopathology when available.

Eligibility:

Histological confirmation of prostate cancer

Age >=18 years old

Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.

Patients must have either:

* Confirmation of prostate cancer with identifiable metastatic disease on at least 1 clinically indicated imaging modality. If there is only soft tissue metastasis, one lesion must measure at least 6 mm or greater. OR
* Documented history of metastatic prostate cancer.

Design:

Two Cohort study

Cohort 1: Stable/Decreasing Prostate Specific Antigen (PSA): PSA must be equal to or less than 0.5 ng/mL value of the last PSA obtained (at least one month apart)

Cohort 2: Rising PSA: PSA must be greater than 0.5 ng/mL above the last PSA value obtained on at least two occasions within 1 year

Patients will undergo DCFPyL PET/CT (or PET/MRI), NaF-PET/CT, and FDG PET/CT within 21 days of each other. The order obtained does not matter.

The DCFPyL PET/CT (or PET/MRI) will be compared with the NaF-PET/CT and FDG PET/CT and standard chest/abdomen/pelvis CT.

DCFPyL PET/CT (or PET/MRI) detection of metastatic disease will be assessed by visual qualitative assessment as positive, equivocal, or negative. Sites of equivocal or positive metastatic disease will have a quantitative PET assessment (SUVmax, SUVmean).

A mandatory research biopsy will be performed under image guidance on a suspicious lesion, if feasible.

The patients will be followed yearly for 4 years by chart review, phone-call, email or any other NIH approved platform for PSA relapse and radiologic evidence of metastatic disease. Additional 18F-DCFPyL and 18F-FDG PET/CTs might be performed during the subject s follow up period there has been a considerable change in patient status (progression or response) based on PSA value, symptomatology, bone scan or CT findings.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Patients must have confirmation of prostate cancer with identifiable metastatic disease on at least 1 clinically indicated imaging modality. If there is only soft tissue metastasis, one lesion must measure at least 6 mm or greater. OR Documented history of metastatic prostate cancer.
* Patients must be co-enrolled on a UOB, GMB or ROB protocol
* Histological confirmation of prostate cancer
* Patients must be willing to undergo mandatory research biopsy

EXCLUSION CRITERIA:

* Subjects for whom participating would significantly delay the scheduled standard of care therapy.
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics
* Other medical conditions deemed by the principal investigator (or associates) to make the subject unsafe/ineligible for protocol procedures.
* Subjects weighing greater than 350 lbs. (weight limit for scanner table), or unable to fit within the imaging gantry
* Serum creatinine greater than 2 times the upper limit of normal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2028-02-06 (Estimated); Study Completion 2028-02-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of DCFPyL-PET/CT diagnostics | 36 months
  Accuracy of DCFPyL-PET/CT diagnostics

SECONDARY OUTCOMES:
PSMA expression in lesion samples from patients with presumed stable disease and actively expanding disease | 36 months
  Correlation between PSMA expression and PSA levels
Association between PSA parameters and the number of metastases identified with DCFPyL- PET/CT (or PET/MRI imaging if available). | 36 months
  Correlation between PSA parameters and the number of metastases identified with DCFPyL- PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Szabo Z, Mena E, Rowe SP, Plyku D, Nidal R, Eisenberger MA, Antonarakis ES, Fan H, Dannals RF, Chen Y, Mease RC, Vranesic M, Bhatnagar A, Sgouros G, Cho SY, Pomper MG. Initial Evaluation of [(18)F]DCFPyL for Prostate-Specific Membrane Antigen (PSMA)-Targeted PET Imaging of Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):565-74. doi: 10.1007/s11307-015-0850-8. PMID 25896814
- [Background] Cho SY, Gage KL, Mease RC, Senthamizhchelvan S, Holt DP, Jeffrey-Kwanisai A, Endres CJ, Dannals RF, Sgouros G, Lodge M, Eisenberger MA, Rodriguez R, Carducci MA, Rojas C, Slusher BS, Kozikowski AP, Pomper MG. Biodistribution, tumor detection, and radiation dosimetry of 18F-DCFBC, a low-molecular-weight inhibitor of prostate-specific membrane antigen, in patients with metastatic prostate cancer. J Nucl Med. 2012 Dec;53(12):1883-91. doi: 10.2967/jnumed.112.104661. PMID 23203246
- [Background] Chen Y, Pullambhatla M, Foss CA, Byun Y, Nimmagadda S, Senthamizhchelvan S, Sgouros G, Mease RC, Pomper MG. 2-(3-1-Carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl-ureido)-pentanedioic acid, [18F]DCFPyL, a PSMA-based PET imaging agent for prostate cancer. Clin Cancer Res. 2011 Dec 15;17(24):7645-53. doi: 10.1158/1078-0432.CCR-11-1357. Epub 2011 Oct 31. PMID 22042970
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0089.html